CLINICAL TRIAL: NCT06964334
Title: The Effect of Vitamin D Supplement as Adjuvant Therapy in Eradication of Helicobacter Pylori Infection
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Samy Abdelsamie Sayed, residant doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: vit D supplement h.pylori
Record Dates: First submitted 2025-05-01; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Lansoprazole; Amoxicillin; Clarithromycin; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Active Comparator): include 35 patients with helicobacter pylori infection with clarithromycin based triple therapy and vitamin D supplement.
  Interventions: Drug: Lansoprazole; Drug: amoxicillin; Drug: clarithromycin; Drug: vitamin D
- Group B (Active Comparator): include 35 patients with helicobacter pylori infection with clarithromycin based triple therapy and without vit D supplement.
  Interventions: Drug: Lansoprazole; Drug: amoxicillin; Drug: clarithromycin

INTERVENTIONS:
Drug: Lansoprazole — oral lansoprazole (1 mg/kg per day, max. 30 mg bid)for 14 day
Drug: amoxicillin — amoxicillin (50 mg/kg per day, max. 1 g bid) for 14 day
Drug: clarithromycin — oral clarithromycin (15 mg/kg per day, max. 500 mg bid) for 14 day
Drug: vitamin D — vitamin D therapy of 4000-5000 units daily in patients over 12 months old.
  Arms: Group A

SUMMARY:
Helicobacter pylori (H. pylori) is one of the most common chronic infections worldwide. The mode of transmission of H. pylori is through the fecal-oral or oral-oral routes.

Chronic gastritis has been linked to helicobacter pylori (H. pylori) infection. Peptic ulcer disease, gastric adenocarcinoma, and gastric lymphoma are all linked to this condition .

In Egypt, a high prevalence of H. pylori infections has been reported, ranging from 70% in the general population , 73% among school children , up to 88% in patients with chronic active HCV .

In 2007, the American College of Gastroenterology estimated that the cure rate for H. pylori infections was 70-85 percent with the use of a proton pump inhibitor (PPI), clarithromycin, and amoxicillin or metronidazole .

children with H. pylori infection do not have severe digestive symptoms. pylori infection represents a key factor in the pathogenesis of duodenal ulcer and chronic gastritis in children. In addition, H. pylori infection has also been reported to have extra-digestive consequences .

A recent comprehensive evaluation found that sequential and conventional triple treatment had a cure rate of 84% .

The infected macrophage is unable to create enough 1,25-(OH)2D to control the synthesis of AMP cathelicidin when it is vitamin D deficient .

vitamin D has a powerful systemic antibacterial impact by enhancing the activity of monocytes and macrophages. Most illnesses seem to benefit from a vitamin D-rich condition .

Vitamin D-deficient subjects might be more prone to developing H. pylori infection .

DETAILED DESCRIPTION:
To assess the efficacy of adding vitamin D supplement as adjuvant therapy in eliminating helicobacter pylori infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 1 to 16 years old who present with helicobacter pylori infection diagnosed by positive stool antigen test for helicobacter pylori infection presented with weight loss, abdominal pain, or failure to surive symptoms for at least 1 month.

Exclusion Criteria:

- 1. Known hypersensitivity to PPIS or antibiotics. 2. Patients who have previously received helicobacter pylori eradication treatment, corticosteroids/immunosuppressive treatment and acid suppressive treatment in the prior 2 months.

3. History of systemic inflammatory or autoimmune disorders, gastric surgery, renal failure, liver cirrhosis and malignancies 4. Abnormal birth history such as premature birth and asphyxia or with severe disease history, such as genetic metabolic disease, congenital dysplasia, feeding difficulties, severe malnutrition, repeated respiratory diseases.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
cure rate after treatment | 3 months
  compare cure rate between two groups